CLINICAL TRIAL: NCT00273403
Title: Outcome Evaluation of Minority AIDS Initiative Programs in the New York EMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The New York Academy of Medicine (Other)
Collaborators: Public Health Solutions (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112299
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2006-09

CONDITIONS: HIV Infections
Keywords: HIV; Minority Groups; Health Services Accessibility; Quality of Life
MeSH Terms: conditions — HIV Infections | interventions — Maintenance; Health Services Accessibility

INTERVENTIONS:
Behavioral: Maintenance in Care Services
Behavioral: Access to Care Services

SUMMARY:
This outcome evaluation effort provides the opportunity to learn what programmatic approaches effectively address two of the most difficult hurdles in HIV health services delivery: (1) getting people who would benefit from health care to use it and (2) getting people who do use health care to do so more consistently and effectively. The New York HIV Planning Council (through MHRA) has funded 23 agencies to achieve these objectives for people of color with HIV disease.

DETAILED DESCRIPTION:
All clients are assessed upon entry into the program, have their service utilization tracked, and then are reassessed at three, six, and twelve months following program entry.

The main client-level data elements collected during baseline and follow-up interviews are the following:

* Biological markers (including HIV status, viral load, t-cell count)
* Demographic characteristics
* Adherence to treatment
* Barriers to care
* Social support
* Substance use and treatment
* Functional health status

Functional Health Status is used in this evaluation as the primary measure of final client "outcomes." The Functional Health Status items we use are from the ACTG SF-21 (a modified version of the Medical Outcomes Study instrument).

The overall evaluation objectives are to:

* Describe the change in functional health status for different populations and groups of clients.
* Identify services or constellations of services and intensity of services associated with change in functional health status.
* Assess whether programs meet intermediate objectives (decreased drug use, increased service use, improved housing stability).
* Identify barriers to access to and maintenance in care.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Not in HIV care, or difficulty being maintained in HIV care
* HIV-negative but at high risk of HIV infection

Exclusion Criteria:

* HIV-negative and not at high risk of HIV infection

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5100
Dates: Start 1999-11; Study Completion 2006-11

PRIMARY OUTCOMES:
Functional Health Status (ACTG SF-21): at 3, 6, and 12 mos.

SECONDARY OUTCOMES:
Housing stability: at 3, 6, and 12 months
Substance use: at 3, 6, and 12 months
Whether receiving HIV primary care: at 3, 6, and 12 months
Whether on HIV meds: at 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Chin, PhD, Principal Investigator — New York Academy of Medicine
Locations (23):
- United States (23):
  - SUNY Downstate Medical Center, Brooklyn, New York
  - HHC Cumberland Diagnostic and Treatment Center, Brooklyn, New York
  - Interfaith Medical Center, Brooklyn, New York
  - Mount Vernon Hospital, Mount Vernon, New York
  - Partnership Homeless Services Corp., New York, New York
  - Betances Health Center, New York, New York
  - Saint Vincents Hospital and Medical Center, New York, New York
  - Bellevue Hospital Center, New York, New York
  - William F. Ryan Community Health Center, New York, New York
  - African Services Committee, New York, New York
  - The Bridge, Inc., New York, New York
  - Settlement Health, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - New York Harm Reducation Educators, Inc., New York, New York
  - Harlem Hospital Center, New York, New York
  - Planned Parenthood of New York City, Project Street Beat, The Bronx, New York
  - Urban Horizons, The Institute for Urban Family Health, The Bronx, New York
  - Health People, The Bronx, New York
  - Bronx Lebanon Hospital Center, The Bronx, New York
  - Health Center at Tremont, North Bronx Healthcare Network, The Bronx, New York
  - Greyston Health Services, Inc., Yonkers, New York
  - Saint Johns Riverside Hospital, Park Care Pavilion (ATC program), Yonkers, New York
  - Saint Johns Riverside Hospital, Park Care Pavilion (MIC Program), Yonkers, New York